CLINICAL TRIAL: NCT00777101
Title: A Phase 2 Randomized Open-Label Study of Neratinib Versus Lapatinib Plus Capecitabine For The Treatment Of ErbB-2 Positive Locally Advanced Or Metastatic Breast Cancer
Brief Title: Study Evaluating Neratinib Versus Lapatinib Plus Capecitabine For ErbB2 Positive Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3144A2-3003 / B1891003
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Results first posted 2017-11-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-07

CONDITIONS: Advanced Breast Cancer; Breast Cancer
Keywords: HER2; ErbB2; metastatic; neratinib; lapatinib; capecitabine; HKI-272; Nerlynx; PB-272
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — neratinib; Lapatinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Neratinib (Experimental)
  Interventions: Drug: Neratinib
- Lapatinib plus Capecitabine (Active Comparator)
  Interventions: Drug: Lapatinib; Drug: Capecitabine

INTERVENTIONS:
Drug: Neratinib — Tablets 240 mg orally once per day until disease progression or unacceptable toxicity
  Other Names: HKI-272
  Arms: Neratinib
Drug: Lapatinib — Tablets 1250 mg orally once per day until disease progression or unacceptable toxicity.
  Other Names: Tykerb, Tyverb
  Arms: Lapatinib plus Capecitabine
Drug: Capecitabine — Tablets 2000 mg/m² given orally in two evenly divided daily doses for first 14 days of each 21 day cycle. Given until disease progression or unacceptable toxicity.
  Other Names: Xeloda
  Arms: Lapatinib plus Capecitabine

SUMMARY:
This is a study of an experimental drug (neratinib) versus a combination of drugs (lapatinib and capecitabine) in women who have erbB-2 (HER-2) positive metastatic or locally advanced breast cancer. The goal of this study is to compare the two regimens in shrinking tumors and extending the lives of women with erbB2 (HER2) positive breast cancer. The study will also compare the safety of the two regimens and to compare quality of life of patients taking the two regimens.

ELIGIBILITY:
Inclusion Criteria:

* Stage IIIB, IIIC, or IV erbB2 (HER2) positive breast cancer
* Prior use of Herceptin (trastuzumab), and a taxane
* Adequate cardiac and renal function

Exclusion Criteria:

* More than 2 prior Herceptin (trastuzumab) regimens or prior use of Xeloda (capecitabine) and / or Tykerb (lapatinib) [Tyverb]
* Bone as the only site of disease
* Active central nervous system metastases (subjects should be stable and off anticonvulsants and steroids)
* Significant gastrointestinal disorder with diarrhea as major symptom

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 233 (Actual)
Dates: Start 2009-02-04 (Actual); Primary Completion 2011-03 (Actual); Study Completion 2018-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Puma, Study Director — Biotechnology
Locations (152):
- United States (44):
  - Arizona Oncology Associates HOPE, Tucson, Arizona
  - Southwest Cancer Care, Murrieta, California
  - UC Irvine Medical Center, Orange, California
  - Aptium Oncology/Comprehensive Cancer Center at Desert Regional Medical Center, Palm Springs, California
  - Redwood Regional Medical Group, Inc., Santa Rosa, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Hematology Oncology Associates, P.C., Stamford, Connecticut
  - Palm Beach Institute of Hematology & Oncology, Boynton Beach, Florida
  - Robert R. Carroll, MD, PA, Gainesville, Florida
  - University of Florida, Jacksonville, Florida
  - Hematology Oncology Associates, Loxahatchee Groves, Florida
  - Mercy Research Institute, Miami, Florida
  - Cancer Centers of Florida, Orlando, Florida
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Cancer Care Specialists Of Central Illinois, Decatur, Illinois
  - Oncology Specialists, SC, Park Ridge, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Central Indiana Cancer Centers, Fishers, Indiana
  - Hematology Oncology of Indiana, Indianapolis, Indiana
  - Floyd Memorial Cancer Center of Indiana, New Albany, Indiana
  - Ashland-Bellefonte Cancer Center, Ashland, Kentucky
  - Owsley Brown Frazier Cancer Center (OBFCC), Louisville, Kentucky
  - Purchase Cancer Group, Paducah, Kentucky
  - Missouri Cancer Associates, Columbia, Missouri
  - Capitol Comprehensive Cancer Care Clinic, Jefferson City, Missouri
  - Arena Oncology Associates, PC, Lake Success, New York
  - Weill Cornell Medical College New York-Presbyterian Hospital Weill, Cornell Breast Center, New York, New York
  - New York Oncology Hematolgy, PC, Troy, New York
  - Oncology Partners Network, Cincinnati, Ohio
  - MetroHealth Medical Center, Cancer Care Center, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center Dept. of Hematology Oncology, Oklahoma City, Oklahoma
  - Northwest Cancer Specialists, PC, Portland, Oregon
  - Lancaster Cancer Center, Lancaster, Pennsylvania
  - Allegheny General Hospital Allegheny Cancer Center, Pittsburgh, Pennsylvania
  - Cookeville Regional Medical Center, Cookeville, Tennessee
  - Center for Biomedical Research, Knoxville, Tennessee
  - Thompson Cancer Survival Center Thompson Oncology Group, Knoxville, Tennessee
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - Texas Oncology, P.A., Austin, Texas
  - El Paso Cancer Treatment Center - West, El Paso, Texas
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - HOPE Oncology, Richardson, Texas
  - Cancer Care Network of South Texas-HOAST, San Antonio, Texas
  - East Texas Medical Center Cancer Institute, Tyler Hematology Oncology, Tyler, Texas
- Australia (4):
  - Mater Private Centre for HOCA, South Brisbane, Queensland
  - Medical Oncology Royal Adelaide Hospital, Adelaide, South Australia
  - Western Hospital, Footscray, Victoria
  - Mount Hospital, West Perth
- AKH Wien Universitaetsklinik fuer Innere Medizin I Klinische Abteilung für Onkologie, Vienna, Austria
- Institut Jules Bordet Unite du Chimiotherapie, Brussels, Belgium
- Bulgaria (3):
  - District Dispensary for Oncology Diseases Internal Unit- Sofia EOOD, Dept. of Chemotherapy, Sofia
  - UMHAT Tzaritza Yoanna, Sofia
  - Interdistrict Dispensary for Oncology Diseases -Internal Unit- Department Oncotherapy and Palliative Care, Varna
- Canada (2):
  - BC Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - Centre Hospitalier Affilie Universitaire de Quebec Hopital du St-Sacrement, Québec, Quebec
- Croatia (3):
  - General Hospital Varazdin, Varaždin
  - University Hospital Center Zagreb, Zagreb
  - University Hospital Sestre Milosrdnice, Zagreb
- Fakultni nemocnice Olomouc Klinika onkologie, Olomouc, Czechia
- France (4):
  - Centre Oscar Lambret Departement de senologie, Lille
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Poitiers Service d'oncologie medicale, Poitiers
  - Institut Gustave ROUSSY Service de Pathologie mammaire, Villejuif
- Germany (2):
  - Universitaetsklinikum Hamburg-Eppendorf Klinik und Poliklinik fuer Gynaekologie, Hamburg
  - Nationales Centrum fuer Tumorerkrankungen Sektion Gynaekologische Onkologie, Heidelberg
- Theagenio Anticancer Hospital of Thessaloniki, Thessaloniki, Greece
- Hong Kong (3):
  - Department of Clinical Oncology, Tuen Mun Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - UNIMED Medical Institute, Comprehensive Centre for Breast Diseases, Hong Kong
- Hungary (6):
  - Fovarosi Onkormanyzat Szent Janos Korhaza es Eszak-budai Egyesitett Korhazai, Onkologia, Budapest
  - Orszagos Onkologiai Intezet "B" Belgyogyaszati osztaly, Budapest
  - Bacs-Kiskun Megyei Korhaz Onkoradiologiai Kozpont, Kecskemét
  - Josa Andras Oktatokorhaz / Onkoradiologiai Osztaly, Nyíregyháza
  - Szegedi Tudomanyegyetem Onkoterapias Klinika, Szeged
  - Hospital of County Veszprem, Veszprém
- Italy (2):
  - Ospedale Misericordia e Dolce c/o UO Oncologia Medica, Prato
  - Istituto Regina Elena, Struttura Complessa Oncologia Medica A, Roma
- Japan (20):
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - National Cancer Center Hospital, Tsukiji, Tokyo
  - Aichi Cancer Center, Aichi
  - Chiba Cancer Center, Chiba
  - National Cancer Center Hospital East, Chiba
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Hiroshima City Hospital, Hiroshima
  - Hyogo Cancer Center, Hyōgo
  - Hakuaikai Medical Corporation Sagara Hospital, Kagoshima
  - Tokai University Hospital, Kanagawa
  - Kumamoto Municipal Hospital, Kumamoto
  - Kyoto University Hospital, Kyoto
  - Niigata Cancer Center Hospital, Niigata
  - National Hospital Organization Osaka National Hospital, Osaka
  - Saitama Cancer Center, Saitama
  - Shizuoka Cancer Center, Shizuoka
  - Jichi Medical University Hospital, Tochigi
  - St. Luke's International Hospital, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research Department of Medical Oncology, Tokyo
  - Tokyo Metropolitan Cancer&Infectious disease Ctr Komagome Hp, Tokyo
- King Hussein Cancer Centre, Amman, Jordan
- Oca Hospital / Monterrey International Research Center, Monterrey, Nuevo León, Mexico
- Poland (4):
  - Bialostockie Centrum Onkologii im. M. Sklodowskiej-Curie w Bialymstoku Specjalistyczny Szpital Onkologiczn, Bialystok
  - Uniwersyteckie Centrum Kliniczne w Gdansku Klinika Onkologii i Radioterapii, Gdansk
  - Szpital Uniwersytecki w Krakowie Oddzial KIiniczny Kliniki Onkologii, Krakow
  - Centrum Onkologii Ziemi Lubelskiej im. SW. Jana z Dukli, Lublin
- Metropolitan Oncology Center, San Juan, PR, Puerto Rico
- Romania (4):
  - Institutul Oncologic "Prof. Dr. Alex. Trestioreanu", Bucharest
  - Spitalul Universitar de Urgenta, Bucharest
  - Centrul de Oncologie Medicala, Iași
  - Spitalul Clinic Judetean, Sibiu
- Russia (9):
  - Scientific Research Institute of Oncology N.N. Petrov, Pesochny, Sankt-Peterburg
  - Russian Oncology Research Centre of RAMS, Moscow
  - GUZ Perm Regional Oncology Dispensary, Perm
  - Ryazan State Medical University I.P.Pavlov of Federal Agency in Healthcare and Social Development, Ryazan
  - SIH Leningrad Regional Oncology Dispensary, Saint Petersburg
  - GUZ City Clinical Oncology Dispensary, Saint Petersburg
  - St. Petersburg State Medical University I.P.Pavlov of Roszdrav, Saint Petersburg
  - SIH Oncology Dispensary # 2 Of Department of Public Health, Sochi
  - Republican Clinical Oncology Dispensary of Ministry of Healthcare of Bashkortostan Republic, Ufa
- Serbia (2):
  - Institute of Oncology and Radiology of Serbia, Belgrade
  - Klinicko Bolnicki Centar (KBC) Bezanijska Kosa (Medical Centre ''Bezanijska Kosa'' (MCBK)), Belgrade
- Johns Hopkins Singapore International Medical Centre, Singapore, Singapore
- Institute for Oncology Department for Medical Oncology, Ljubljana, Slovenia
- South Africa (4):
  - The Medical Oncology Centre of Rosebank, Johannesburg, Gauteng
  - Eastleigh Breast Care Centre, Lynnwood, Gauteng
  - Hopelands Oncology Centre, Durban, KwaZulu-Natal
  - GVI Oncology Trial Unit Room 110 Panorama Medical Centre, Kraaifontein, Western Cape
- South Korea (4):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Samsung Medical Center, Seoul, Korea
  - Yonsei University Health System - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (15):
  - Hospital Germans Trias i Pujol Servicio de Oncologia, Badalona, Barcelona
  - Corporacio Sanitaria Parc Tauli Servicio de Oncologia, Sabadell, Barcelona
  - Hospital Mutua de Terrassa Servicio de Oncologia, Terrassa, Barcelona
  - Hospital Central de Asturias Servicio de Oncologia, Planta Baja Oeste, Edificio Principal, Oviedo, Principality of Asturias
  - Complejo Hospitalario U. de A Coruña Hospital Teresa Herrera Servicio de Oncologia, A Coruña
  - Hospital General Universitario de Alicante Servicio de Oncologia, Alicante
  - Hospital San Pedro de Alcantara Servicio de Oncologia, Cáceres
  - Hospital Provincial (Reina Sofia) Servicio de Oncologia, Córdoba
  - Hospital Universitario Dr. Josep Trueta Servicio de Oncologia, Girona
  - Centro Hospitalario de Jaen Servicio de Oncologia, Jaén
  - Hospital Gregorio Marañon Servicio de Oncologia, Madrid
  - Centro Oncologico M.D. Anderson Internacional, Madrid
  - Instituto Valenciano de Oncologia Servicio de Oncologia, Valencia
  - Hospital Clinico Universitario de Valencia Servicio de Hematologia y Oncologia, Valencia
  - Hospital Universitario Miguel Servet Servicio de Oncologia, Zaragoza
- Switzerland (3):
  - University of Lausanne Hospitals CHUV, Lausanne
  - Kantonsspital Winterthur Medizinische Onkologie, Winterthur
  - Abteilung fuer Onkologie Departement für Innere, Zurich
- National Taiwan University Hospital, Taipei, Taiwan
- Division of Medical Oncology, Department of Medicine, Bangkok Noi, Bangkok, Thailand
- United Kingdom (3):
  - Broomfield Hospital, Chelmsford, Essex
  - Royal Marsden NHS Foundation Trust & Institute of Cancer Research, London
  - The Royal Marsden NHS Foundation Trust & Institute of Cancer Research, London

REFERENCES:
- [Derived] Martin M, Bonneterre J, Geyer CE Jr, Ito Y, Ro J, Lang I, Kim SB, Germa C, Vermette J, Wang K, Wang K, Awada A. A phase two randomised trial of neratinib monotherapy versus lapatinib plus capecitabine combination therapy in patients with HER2+ advanced breast cancer. Eur J Cancer. 2013 Dec;49(18):3763-72. doi: 10.1016/j.ejca.2013.07.142. Epub 2013 Aug 15. PMID 23953056

RESULTS

PARTICIPANT FLOW:
Groups:
- Neratinib: Neratinib
  Neratinib: Tablets, 240mg once per day until disease progression or unacceptable toxicity
- Lapatinib+Capecitabine: Lapatinib plus Capecitabine
  Lapatinib: Tablets 1250mg once per day until disease progression or unacceptable toxicity.
  Capecitabine: Tablets 2000mg/m2 given in two evenly divided daily doses for first 14 days of each 21 day cycle. Given until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Neratinib | Lapatinib+Capecitabine
Started | 117 | 116
Treated | 116 | 115
Completed | 55 | 65
Not Completed | 62 | 51
Not completed — Death | 48 | 43
Not completed — Withdrawal by Subject | 11 | 6
Not completed — Lost to Follow-up | 2 | 1
Not completed — Discontinuation of Study by Sponsor | 1 | 0
Not completed — Failed to Return | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Neratinib | Lapatinib+Capecitabine | Total
Number analyzed (Participants) | 117 | 116 | 233
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 104 | 100 | 204
  >=65 years | 13 | 16 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (10.11) | 54.7 (13.8) | 54.3 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 116 | 233
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 32 | 46 | 78
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 77 | 64 | 141
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression Free Survival, Measured in Months, for Subjects Randomized. Investigator assessment. The time interval from the date of randomization until the earliest date of progression per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) or death due to any cause. For subjects without death or progression, censorship was at the last valid tumor assessment.
Time Frame: From randomization date to progression or death, assessed up to 69 months
Population: Intent to Treat population, includes all subjects who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Neratinib | Lapatinib+Capecitabine
Number analyzed (Participants) | 117 | 116
months | 4.53 [3.12 to 5.65] | 6.83 [5.85 to 8.21]
Statistical Analysis 1: Comparison: Neratinib vs Lapatinib+Capecitabine; Test type: Non-Inferiority — Non-inferiority of neratinib vs lapatinib + capecitabine was to be concluded if the upper limit of the 95% confidence interval (CI) for the hazard ratio was 1.15 or less; p = 0.231, Log Rank; The log-rank test comparing treatment groups is stratified by region; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.89 to 1.60] — The hazard ratio is estimated by stratified Cox model. The Cox model is stratified by region

2. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was defined as the time from randomization to death due to any cause. Subjects last known to be alive were censored at the last date of last contact or the data cutoff employed for the analysis, whichever was earlier.
Time Frame: From randomization date to death, assessed up to 69 months
Population: Intent to Treat population, includes all subjects who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Neratinib | Lapatinib+Capecitabine
Number analyzed (Participants) | 117 | 116
months | 19.74 [18.20 to NA] — Insufficient number of participants to calculate the upper bound of the confidence interval. | 23.62 [18.00 to NA] — Insufficient number of participants to calculate the upper bound of the confidence interval.

3. Secondary Outcome: Objective Response Rate (ORR).
Description: Objective Response Rate, investigator assessment. The ORR was defined as the percentage of participants demonstrating a confirmed objective response, either Complete Response (CR) or Partial Response (PR) during the study per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v.1.0: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; and Non-PD for non-target lesions, and no new lesions.
Time Frame: From randomization date to progression or last tumor assessment, assessed up to 69 months
Population: Intent to Treat population, includes all subjects who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neratinib | Lapatinib+Capecitabine
Number analyzed (Participants) | 117 | 116
percentage of participants | 29.1 [21 to 38.2] | 40.5 [31.5 to 50.0]

4. Secondary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate (CR, PR, or SD = 24 weeks) for women For ErbB2 Positive Advanced Breast Cancer. Clinical benefit rate was the percentage of subjects who achieved overall tumor response per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.0: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
  Clinical Benefit (CB) = CR + PR + SD >= 24 weeks.
Time Frame: From randomization date to progression or last tumor assessment, assessed up to 69 months
Population: Intent to Treat population, includes all subjects who were randomized.
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neratinib | Lapatinib+Capecitabine
Number analyzed (Participants) | 117 | 116
percentage of participants | 44.4 [35.3 to 53.9] | 63.8 [54.4 to 72.5]

5. Secondary Outcome: Duration of Response
Description: Duration of response was measured from the time at which response criteria were met for complete response (CR) or partial response (PR) (whichever status was recorded first) until the first date of recurrence or progressive disease (PD) or death. For subjects without death or progression, censorship was at the last valid tumor assessment per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.0: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: From start date of response to first PD, assessed up to 69 months after the first subject was randomized.
Population: No. of Subjects with either complete or partial response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Neratinib | Lapatinib+Capecitabine
Number analyzed (Participants) | 34 | 47
months | 12.48 [8.31 to 14.75] | 7.98 [5.49 to 11.76]

6. Secondary Outcome: Frequency of CNS Metastases (Frequency)
Description: The percent of patients with symptomatic or progressive CNS lesions was the proportion of subjects who had PD considering CNS lesions only, according to RECIST criteria.
Time Frame: From randomization date to first CNS symptom or lesions
Population: Intent to Treat population, includes all subjects who were randomized.
Measure: Number; unit: percentage of participants
Groups:
- Lapatinib+Capecitabine: Lapatinib+Capecitabine
  Lapatinib: Tablets 1250mg once per day until disease progression or unacceptable toxicity.
  Capecitabine: Tablets 2000mg/m2 given in two evenly divided daily doses for first 14 days of each 21 day cycle. Given until disease progression or unacceptable toxicity.
Arm/Group | Neratinib | Lapatinib+Capecitabine
Number analyzed (Participants) | 117 | 116
percentage of participants | 9.4 | 12.9

7. Secondary Outcome: Time to CNS Metastases
Description: Time to symptomatic or progressive Central nervous system (CNS) lesions. Time to symptomatic or progressive CNS lesions was the time from the date of randomization until the date of progressive disease (PD) considering CNS lesions only (ie, appearance of newly diagnosed CNS lesions or progressive CNS lesions).
Time Frame: From randomization date to first CNS symptom or lesions
Population: Intent to Treat population, includes all subjects who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Neratinib | Lapatinib+Capecitabine
Number analyzed (Participants) | 117 | 116
months | 19.68 [19.68 to 20.99] | NA [NA to NA] — Insufficient number of participants with events to calculate the median and confidence intervals.

ADVERSE EVENTS:
Time Frame: From First Dose through 28 days after last dose, assessed up to 69 months.
Description: See below
Arm/Group | Neratinib | Lapatinib+Capecitabine
Serious Adverse Events (participants affected / at risk) | 31/116 | 24/115
Other Adverse Events (participants affected / at risk) | 113/116 | 114/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neratinib (N=116) | Lapatinib+Capecitabine (N=115)
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 4
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 3
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 3
Asthenia (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Disease progression (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 2
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 3
Sudden death (General disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Mastitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Wound sepsis (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain oedema (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 0 | 2
Encephalopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 1
Subclavian artery stenosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neratinib (N=116) | Lapatinib+Capecitabine (N=115)
Anaemia (Blood and lymphatic system disorders) | 9 | 5
Leukopenia (Blood and lymphatic system disorders) | 5 | 12
Neutropenia (Blood and lymphatic system disorders) | 5 | 17
Abdominal pain (Gastrointestinal disorders) | 11 | 14
Abdominal pain upper (Gastrointestinal disorders) | 8 | 12
Constipation (Gastrointestinal disorders) | 8 | 12
Diarrhoea (Gastrointestinal disorders) | 100 | 82
Dyspepsia (Gastrointestinal disorders) | 13 | 11
Nausea (Gastrointestinal disorders) | 50 | 48
Stomatitis (Gastrointestinal disorders) | 9 | 28
Vomiting (Gastrointestinal disorders) | 38 | 25
Asthenia (General disorders) | 22 | 13
Fatigue (General disorders) | 30 | 30
Influenza like illness (General disorders) | 4 | 6
Mucosal inflammation (General disorders) | 6 | 19
Pain (General disorders) | 7 | 8
Pyrexia (General disorders) | 6 | 10
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 | 27
Cystitis (Infections and infestations) | 7 | 5
Nasopharyngitis (Infections and infestations) | 3 | 10
Paronychia (Infections and infestations) | 6 | 24
Upper respiratory tract infection (Infections and infestations) | 6 | 5
Urinary tract infection (Infections and infestations) | 6 | 10
Alanine aminotransferase increased (Investigations) | 11 | 15
Aspartate aminotransferase increased (Investigations) | 10 | 19
Blood alkaline phosphatase increased (Investigations) | 8 | 4
Blood bilirubin increased (Investigations) | 0 | 6
Weight decreased (Investigations) | 15 | 13
Decreased appetite (Metabolism and nutrition disorders) | 33 | 23
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 6 | 0
Dizziness (Nervous system disorders) | 6 | 13
Dysgeusia (Nervous system disorders) | 4 | 8
Headache (Nervous system disorders) | 24 | 12
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 10
Insomnia (Psychiatric disorders) | 9 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 10
Acne (Skin and subcutaneous tissue disorders) | 3 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 10
Nail disorder (Skin and subcutaneous tissue disorders) | 3 | 13
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 9 | 77
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 17
Rash (Skin and subcutaneous tissue disorders) | 26 | 41
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 6
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 12

LIMITATIONS AND CAVEATS:
Pharmacokinetic Analyses not included here; they are part of a population PK analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less